CLINICAL TRIAL: NCT01792830
Title: Prospective Study Aim to Determine the Efficacy and Safety of a Glargine-based Hospital Discharge Algorithm in Cardiac Surgery Patients With Perioperative Hyperglycemia
Brief Title: Efficacy and Safety of a Glargine-based Hospital Discharge Algorithm in Coronary Artery Bypass Graft (CABG) Patients
Acronym: CABG-D/C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056365
Record Dates: First submitted 2012-08-14; First posted 2013-02-15 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Poor Glycemic Control
Keywords: Coronary Artery Bypass Graft surgery
MeSH Terms: interventions — Metformin; Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Control HbA1c < 7% (No Intervention): Subjects not requiring coronary artery bypass graft surgery (CABG), with no history of diabetes with HbA1c <7% not requiring subcutaneous insulin in the hospital will be discharged on no antidiabetic therapy.
- Diabetic/ Metformin and 50-Glargine HbA1c 7%- 9% (Active Comparator): Subjects requiring coronary artery bypass graft surgery (CABG) with a history of diabetes with HbA1c between 7% and 9% requiring subcutaneous insulin therapy in the hospital will be discharged on oral metformin and a single dose of basal (glargine) insulin at 50% of total daily hospital dose.
  Interventions: Drug: Metformin; Drug: Glargine insulin
- Diabetic/ Metformin and 80-Glargine HbA1c 7%-9%% (Active Comparator): Subjects requiring coronary artery bypass graft surgery (CABG) with a history of diabetes with HbA1c 7%- 9% will be discharged on oral metformin and a single dose of basal (glargine) insulin at 80% of total daily hospital dose or with basal bolus regimen at same inpatient total daily insulin dose.
  Interventions: Drug: Metformin; Drug: Glargine insulin
- No diabetes/ Metformin only (Active Comparator): Subjects requiring coronary artery bypass graft surgery (CABG) with no history of diabetes with HbA1c <7% and persistent hyperglycemia requiring subcutaneous (SC) insulin therapy in the hospital will be discharged on oral metformin.
  Interventions: Drug: Metformin
- Diabetic/antidiabetic regimen (Active Comparator): Subjects requiring coronary artery bypass graft surgery (CABG) with a history of diabetes with HbA1c <7% will be discharged on their same outpatient antidiabetic regimen. Subjects will receive one of the three treatment options based on their blood glucose levels: Metformin alone, both metformin and glargine insulin or glargine alone.
  Interventions: Drug: Metformin; Drug: Glargine insulin
- No diabetes/ Insulin only (Active Comparator): Subjects requiring coronary artery bypass graft surgery (CABG) with no history of diabetes with HbA1c <7% and persistent hyperglycemia will be given subcutaneous (SC) insulin therapy in the hospital.
  Interventions: Drug: Glargine insulin
- Diabetes/Insulin only (Active Comparator): Subjects requiring coronary artery bypass graft surgery (CABG) with an admission HbA1c >9% and persistent hyperglycemia will be given basal insulin (glargine) once daily, at the same time of the day and rapid-acting insulin (glulisine) before meals.
  Interventions: Drug: Glargine insulin; Drug: Glulisine

INTERVENTIONS:
Drug: Metformin — Metformin is an oral antidiabetic agent used to control high blood glucose levels and is given in divided doses with meals. During treatment initiation and dose titration, the patient's blood glucose levels will be used to determine the therapeutic response to metformin and identify the minimum effective dose for the patient.
  Patients without a history of diabetes and admission HbA1c < 7% requiring SC insulin therapy in the hospital will be discharged on metformin monotherapy.
  Treatment naïve patients with an HbA1c between 7% and 9% prior to admission will be discharged on metformin monotherapy or a combination of metformin and a single dose of subcutaneous insulin.
  Other Names: Glucophage
  Arms: Diabetic/ Metformin and 50-Glargine HbA1c 7%- 9%; Diabetic/ Metformin and 80-Glargine HbA1c 7%-9%%; Diabetic/antidiabetic regimen; No diabetes/ Metformin only
Drug: Glargine insulin — Glargine is a recombinant human insulin analog that exhibits a constant glucose-lowering profile over 24 hours and permits once-daily dosing. It is administered subcutaneously once a day at the same time every day.
  Patients with an HbA1c between 7% and 9% requiring subcutaneous insulin therapy in the hospital will be discharged on oral metformin and a single dose of glargine insulin at 50% of total daily hospital dose.
  Patients with an HbA1c > 9% will be discharged on oral metformin and a single dose of glargine insulin at 80% of total daily hospital dose.
  Other Names: Lantus
  Arms: Diabetes/Insulin only; Diabetic/ Metformin and 50-Glargine HbA1c 7%- 9%; Diabetic/ Metformin and 80-Glargine HbA1c 7%-9%%; Diabetic/antidiabetic regimen; No diabetes/ Insulin only
Drug: Glulisine — Glulisine is an injectable, recombinant insulin analog. The total daily dose varies between 0.5 to 1 unit/kg/day depending on the levels of blood glucose. Glulisine will be given within 15 minutes before a meal or within 20 minutes after starting a meal.
  Other Names: Apidra
  Arms: Diabetes/Insulin only

SUMMARY:
Most coronary artery bypass graft surgery (CABG) patients develop high blood sugar while they are in the hospital. No studies have shown what the best insulin regimen is for CABG patients with type 2 diabetes is after going home from the hospital. Patients with high blood sugar and diabetes after cardiac bypass surgery will be followed for 3 months to look at how well their treatment(s) for diabetes work after discharge. Patients with diabetes will be discharged on oral antidiabetic drugs or with insulin glargine injections based on their sugar control. Patients with admission HbA1c < 7% (a laboratory value that shows the average blood sugar level in the body over 3 months) will be discharged on the same diabetes medications that they used before coming to the hospital. Those with an HbA1c between 7% and 9% will be discharged on insulin glargine at 50%-80% of the dose used in the hospital and oral antidiabetic drugs. Those with an HbA1c > 9% will be discharged on glargine at 80-100% of the dose used in the hospital in addition to oral antidiabetic drugs or with insulin glargine and insulin glulisine. The primary outcome will be a change in HbA1c at 4 and 12 weeks after discharge.

DETAILED DESCRIPTION:
Hospital discharge represents a critical time for ensuring a safe transition to the outpatient setting and reducing the need for emergency department visits and re-hospitalization. Poor coordination of patient care and education on insulin administration at the time of patient discharge to home may be associated with medical errors that may increase risk of hypoglycemia, hyperglycemia and hospital readmission. No prospective studies have examined the impact of a discharge treatment regimen after cardiac surgery. Therefore, this study aims to determine the efficacy and safety of an HbA1c based treatment algorithm in controlling blood glucose (BG) after discharge. The total duration of the study is 3 months.

This study will include diabetic and non-diabetic subjects who participated in the American Diabetes Association (ADA) trial entitled "Intensive Insulin Therapy in Patients Undergoing Coronary Artery Bypass Surgery." The ADA study is a two-arm randomized multicenter, open-label controlled trial aimed to determine if intensive insulin control with a BG target of 100-140mg/dl will reduce perioperative complications compared to a conventional BG control with a target of 141-180 mg/dl in hyperglycemic subjects who undergo coronary artery bypass graft surgery (CABG).

Treatment recommendations at discharge:

* Patients with admission HbA1c < 7%:

  * Patients without a history of diabetes not requiring subcutaneous (SC) insulin in the hospital will be discharged on no antidiabetic therapy.
  * Patients without a history of diabetes requiring SC insulin therapy in the hospital will be discharged on metformin monotherapy. A patient without a history of diabetes who requires SC insulin is likely a newly diagnosed diabetic. The HbA1c value will be important to confirm the diagnosis. If the HbA1c is >6.5%, he/she will be diagnosed with diabetes. We do not anticipate that a patient without a history of diabetes and with an HbA1c <6.5% will require insulin treatment or oral agents long-term. Those patients will be discharged on no anti diabetic therapy with repeated testing after discharge to rule out diabetes.
  * Patients with a history of diabetes will be discharged on their same outpatient antidiabetic regimen (diet, oral antidiabetic agents and/or insulin).
  * Assure there are no contraindications to oral agents (i.e.Thiazolidinediones (TZDs) and heart failure; metformin and renal failure or heart failure).
* Patients with Admission HbA1c between 7% and 9%:

  * Treatment naïve patients not on any pharmacologic treatment prior to admission will be discharged on metformin monotherapy or a combination of metformin and a single dose of basal (glargine) insulin at 50% of total daily hospital dose.
  * Patients treated with oral antidiabetic agents or glucagon-like peptide-1 (GLP1) analogs prior to admission will be discharged on pre-admission oral antidiabetic therapy plus a single dose of glargine insulin at 50% of the total daily hospital dose.
  * Patients treated with combination of oral antidiabetic agents and basal insulin (NPH insulin also known as Neutral Protamine Hagedorn insulin, glargine, detemir) prior to admission will be discharged on pre-admission oral antidiabetic therapy plus a single dose of glargine insulin or with basal bolus insulin regimen at 50% of total daily hospital dose.
  * Patients not to be treated with oral agents will be discharged on glargine monotherapy or basal bolus at 100% of inpatient total daily dose.
  * Admission HbA1c ≥ 9% prior to admission:
  * Discharge on basal bolus regimen at same inpatient total daily insulin dose.
  * Basal insulin (glargine) once daily, at the same time of the day.
  * Rapid-acting insulin (glulisine) before meals.
  * Alternative treatment: If no contraindications to oral agents (i.e., Thiazolidinediones (TZDs) and heart failure; metformin and renal failure) restart oral agents in combination to glargine once daily at 80% of total daily hospital dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years undergoing primary coronary artery bypass graft surgery (CABG).
2. Post surgical hyperglycemia (Blood glucose >140 mg/dl)
3. Patients with and without a history of type 2 diabetes

Exclusion Criteria:

1. Patients with severely impaired renal function (serum creatinine ≥3.0 mg/dl or a glomerular filtration rate < 30 ml/min) or clinically significant hepatic failure.
2. Subjects with acute hyperglycemic crises such as diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic states.
3. Moribund patients and those at imminent risk of death (brain death or cardiac standstill).
4. Patients or next-to-kin with mental conditions rendering the subject or family member unable to understand the nature, scope, and possible consequences of the study.
5. Female subjects who are pregnant or breast-feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Midtown Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital, Emory University Hospital - Midtown, and Grady Memorial Hospital, in Atlanta, Georgia, from October 2012 to February 2014. Study arms for results are presented to precisely reflect the medication used post-hospital discharge, as prescribed by the participant's provider.
Groups:
- Control, Non-diabetic, no Treatment: Participants who did not have coronary artery bypass graft surgery (CABG), with no history of diabetes and with HbA1C <7%, who did not require subcutaneous insulin in the hospital and were discharged with no antidiabetic therapy.
- Non-diabetic, Metformin: Participants without a history of diabetes and with HbA1C <7%, who were discharged on oral metformin following CABG surgery.
- Non-diabetic, Insulin: Participants without a history of diabetes and with HbA1C< 7% and persistent hyperglycemia requiring subcutaneous insulin therapy in the hospital who were discharged without oral diabetes medication, following CABG surgery.
- Diabetic, HbA1C <7%, Metformin: Participants with a history of diabetes and with HbA1C <7% who were discharged on oral metformin, following CABG surgery.
- Diabetic, HbA1C <7%, Metformin and Insulin Glargine: Participants with a history of diabetes and with HbA1C <7% who were discharged on metformin and insulin glargine, following CABG surgery.
- Diabetic, HbA1C <7%, Insulin Glargine: Participants with a history of diabetes and with HbA1C <7% who were discharged on glargine insulin (a long-acting basal insulin analogue), following CABG surgery.
- Diabetic, HbA1C 7%- 9%, Metformin: Participants with a history of diabetes and with HbA1C between 7% and 9% who were discharged on oral metformin, following CABG surgery.
- Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine: Participants with a history of diabetes and with HbA1C between 7% and 9% who were discharged on oral metformin plus a single dose of glargine insulin or with basal bolus insulin regimen at 50% of total daily hospital dose, following CABG surgery.
- Diabetic, HbA1C 7%-9%, Insulin Glargine: Participants with a history of diabetes and with HbA1C between 7% and 9% who were discharged on glargine insulin (a long-acting basal insulin analogue), following CABG surgery.
- Diabetic, HbA1C >9%, Metformin and Insulin Glargine: Participants with a history of diabetes and with HbA1C >9% who were discharged on oral metformin and glargine insulin to be taken daily at the same time of day or a basal bolus insulin regimen, following CABG surgery.
- Diabetic, HbA1C >9%, Insulin Glulisine: Participants with a history of diabetes and with HbA1C >9% who were discharged on glulisine, a rapid-acting insulin to be taken before meals, following CABG.
Period: Overall Study
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
Started | 84 | 3 | 4 | 21 | 2 | 4 | 14 | 7 | 20 | 4 | 12
Completed (Participants who died in the hospital, before follow-up, are considered as not completing the study.) | 59 | 3 | 4 | 18 | 1 | 3 | 12 | 6 | 11 | 4 | 9
Not Completed | 25 | 0 | 0 | 3 | 1 | 1 | 2 | 1 | 9 | 0 | 3
Not completed — Withdrawal by Subject | 22 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 7 | 0 | 2
Not completed — Death | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine | Total
Number analyzed (Participants) | 84 | 3 | 4 | 21 | 2 | 4 | 14 | 7 | 20 | 4 | 12 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 0 | 1 | 11 | 0 | 1 | 5 | 2 | 8 | 4 | 11 | 84
  >=65 years | 43 | 3 | 3 | 10 | 2 | 3 | 9 | 5 | 12 | 0 | 1 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 0 | 1 | 6 | 1 | 1 | 5 | 1 | 5 | 3 | 3 | 49
  Male | 61 | 3 | 3 | 15 | 1 | 3 | 9 | 6 | 15 | 1 | 9 | 126
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 84 | 3 | 4 | 21 | 2 | 4 | 14 | 7 | 20 | 4 | 12 | 175

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Measured by a Change in HbA1c Levels
Description: Change in the level of HbA1c in a one month period after discharge from the hospital. The A1c test result is reported as a percentage. Higher percentages indicate higher blood glucose levels in the previous three months. A normal HbA1c level is below 5.7 percent.
Time Frame: One month after hospital discharge
Population: This analysis includes participants who had blood drawn one month after hospital discharge. Most patients that completed the discharge part did so over the phone. The "diabetic, HbA1C <7%, metformin and insulin glargine" is not included in this table as no participants in this group had blood drawn for this analysis.
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
Number analyzed (Participants) | 24 | 1 | 2 | 9 | 3 | 6 | 4 | 9 | 3 | 5
percent of glycosylated hemoglobin | 5.09 (0.43) | 5.2 (0.00) | 5.5 (0.5) | 5.8 (0.5) | 6.9 (1.60) | 6.1 (2.60) | 6.3 (0.89) | 6.6 (0.70) | 8.6 (1.9) | 6.9 (0.4)

2. Secondary Outcome: Number of Participants Readmitted to the Hospital
Description: The number of participants that were readmitted to the hospital 3 months after initial hospital discharge
Time Frame: 3 months after discharge
Population: This analysis includes participants who completed the month 3 study visit either in person or by phone.
Measure: Number; unit: participants
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
Number analyzed (Participants) | 41 | 2 | 4 | 3 | 1 | 1 | 6 | 5 | 8 | 3 | 4
participants | 11 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: The Number of Participants Experiencing a Hypoglycemic Event
Description: The number of participants that experienced hypoglycemia, defined as blood glucose levels ≤70 mg/dl.
Time Frame: 3 months after discharge
Population: This analysis includes participants who completed the month 3 study visit either in person or by phone.
Measure: Count of Participants; unit: Participants
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
Number analyzed (Participants) | 41 | 2 | 4 | 3 | 1 | 1 | 6 | 5 | 8 | 3 | 4
Participants | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1

4. Secondary Outcome: The Number of Participants Experiencing a Severe Hypoglycemic Event
Description: The number of participants that experienced severe hypoglycemia, defined as blood glucose levels ≤ 40 mg/dl.
Time Frame: 3 months after discharge
Population: Participants who completed the Month 3 study visit in person or by phone.
Measure: Count of Participants; unit: Participants
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
Number analyzed (Participants) | 41 | 2 | 4 | 3 | 1 | 1 | 6 | 5 | 8 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing a Hyperglycemic Event
Description: The number of participants that experienced hyperglycemia, defined as blood glucose levels ≥ 140 mg/dl.
Time Frame: 3 months after discharge
Population: Participants who completed the Month 3 study visit, in person or by phone.
Measure: Count of Participants; unit: Participants
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
Number analyzed (Participants) | 41 | 2 | 4 | 3 | 1 | 1 | 6 | 5 | 8 | 3 | 4
Participants | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 1 | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a participant signed the consent form until one month after hospital discharge.
Description: Mortality data includes participants who died prior to initial hospital discharge plus those who died during the study follow-up period. Any post-operative complications (including infections and wound infections) are captured as adverse events.
Arm/Group | Control, Non-diabetic, no Treatment | Non-diabetic, Metformin | Non-diabetic, Insulin | Diabetic, HbA1C <7%, Metformin | Diabetic, HbA1C <7%, Metformin and Insulin Glargine | Diabetic, HbA1C <7%, Insulin Glargine | Diabetic, HbA1C 7%- 9%, Metformin | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine | Diabetic, HbA1C 7%-9%, Insulin Glargine | Diabetic, HbA1C >9%, Metformin and Insulin Glargine | Diabetic, HbA1C >9%, Insulin Glulisine
All-Cause Mortality (participants affected / at risk) | 5/84 | 0/3 | 1/4 | 0/21 | 0/2 | 0/4 | 1/12 | 0/7 | 2/20 | 0/4 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/84 | 0/3 | 0/4 | 0/21 | 0/2 | 0/4 | 2/14 | 0/7 | 0/20 | 1/4 | 0/12
Other Adverse Events (participants affected / at risk) | 6/84 | 1/3 | 0/4 | 1/21 | 0/2 | 1/4 | 0/14 | 0/7 | 0/20 | 2/4 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control, Non-diabetic, no Treatment (N=84) | Non-diabetic, Metformin (N=3) | Non-diabetic, Insulin (N=4) | Diabetic, HbA1C <7%, Metformin (N=21) | Diabetic, HbA1C <7%, Metformin and Insulin Glargine (N=2) | Diabetic, HbA1C <7%, Insulin Glargine (N=4) | Diabetic, HbA1C 7%- 9%, Metformin (N=14) | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine (N=7) | Diabetic, HbA1C 7%-9%, Insulin Glargine (N=20) | Diabetic, HbA1C >9%, Metformin and Insulin Glargine (N=4) | Diabetic, HbA1C >9%, Insulin Glulisine (N=12)
Cardiac disorder resulting in inpatient death (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Cardiac disorder resulting in death during hospital readmission (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control, Non-diabetic, no Treatment (N=84) | Non-diabetic, Metformin (N=3) | Non-diabetic, Insulin (N=4) | Diabetic, HbA1C <7%, Metformin (N=21) | Diabetic, HbA1C <7%, Metformin and Insulin Glargine (N=2) | Diabetic, HbA1C <7%, Insulin Glargine (N=4) | Diabetic, HbA1C 7%- 9%, Metformin (N=14) | Diabetic, HbA1C 7%-9%, Metformin and Insulin Glargine (N=7) | Diabetic, HbA1C 7%-9%, Insulin Glargine (N=20) | Diabetic, HbA1C >9%, Metformin and Insulin Glargine (N=4) | Diabetic, HbA1C >9%, Insulin Glulisine (N=12)
Trauma from car accident (Social circumstances) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hematoma (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomach virus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bladder cancer (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Necrotic ulcer (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystectomy (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study had participants from other states who lived more than 50 miles away from the hospitals and did not return for their post-operative care or 12 week follow up. Some subjects preferred to complete follow ups via phone and no blood was drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes